CLINICAL TRIAL: NCT01614275
Title: Using Technology to Expand and Enhance Applied Behavioral Analysis Programs for Children With Autism in Military Families
Brief Title: Using Web-based Technology to Expand and Enhance Applied Behavioral Analysis Programs for Children With Autism in Military Families
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Nebraska (Other)
Collaborators: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Wayne Fisher, Director, Center for Autism Spectrum Disorders, University of Nebraska
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 059-11; W81XWH-11-1-0444 (Other Grant/Funding Number: US ARMY MEDICAL RESEARCH AND MATERIAL COMMAND)
Record Dates: First submitted 2012-06-05; First posted 2012-06-07 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Autism Spectrum Disorders
Keywords: Autism; Early Intervention; Parent Training; EIBI; Applied Behavior Analysis
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Technology-enhanced Parent Training (Experimental): The investigators will demonstrate that web-based instructional technologies provides an efficient and effective mechanism for training military parents of children with autism, regardless of their geographic location, to implement effective behavior management and teaching strategies with high procedural integrity (90% accuracy).
  Interventions: Behavioral: Technology-Enhanced Parent Training
- Technology-enhanced Tutor Training (Experimental): The investigators will demonstrate that web-based instructional technologies provides an efficient and effective mechanism for training tutors to implement early intervention services that are commonly used with children diagnosed with autism with high procedural integrity (above 80%).
  Interventions: Behavioral: Technology-Enhanced Tutor Training
- Technology-enhanced Early Intensive Behavioral Intervention (Experimental): The investigators will demonstrate that technology-enhanced service delivery will provide remote access to efficient and effective EIBI services to military families affected by autism.
  Interventions: Behavioral: Technology-enhanced Early Intensive Behavioral Intervention
- Wait-list No-intervention Control Group (Placebo Comparator): Tutors and families will be assigned to treatment and control groups using the process of minimization, which has been recommended for small clinical trials because it minimizes differences between the groups on relevant covariables while guarding against bias in ways comparable to simple randomization. The control group will not receive intervention services.
  Interventions: Behavioral: No-Intervention

INTERVENTIONS:
Behavioral: Technology-Enhanced Parent Training — The training for the parents of children with autism assigned to the EIBI group will begin with completion of a structured parent-training program for 6 weeks that includes 16 to 18 sessions (three, 90-minute sessions per week). When a new topic is introduced, the initial training will include viewing a Power Point presentation, with embedded video and audio, that explains, in laymen's terms, the basic principles and processes related to the topic. The second part of the training involves a parent recruiting an adult friend, who will play the role of a child with autism. The adult playing the child with autism will wear a Bluetooth earpiece connected to a computer, which in turn will be connected to a UNMC expert. The expert will guide the actions of the adult playing the role of the child such that this confederate "child" will exhibit a variety of target behaviors relevant to the target skill, which will provide an opportunity for immediate feedback.
  Arms: Technology-enhanced Parent Training
Behavioral: Technology-Enhanced Tutor Training — The training for the tutors to work with children diagnosed with autism, who were assigned to the EIBI group, will complete a 40-hour structured training program for 4 to 8 weeks that includes approximately 32 sessions. When a new topic is introduced, the initial training will include viewing a PowerPoint presentation, with embedded video and audio, that explains, in laymen's terms, the basic principles and processes related to the topic. The second part of the training involves a tutor recruiting an adult friend, who will play the role of a child with autism. The adult playing the child with autism will wear a Bluetooth earpiece connected to a computer, which in turn will be connected to a UNMC expert. The expert will guide the actions of the adult playing the role of the child such that this confederate "child" will exhibit a variety of target behaviors relevant to the target skill, which will provide an opportunity for immediate feedback.
  Arms: Technology-enhanced Tutor Training
Behavioral: Technology-enhanced Early Intensive Behavioral Intervention — After training, the ABA tutor and parents will assist in the implementation of early intervention services that will be tailored to the particular needs of the family's child. These programs could include conducting a paired-stimulus preference assessment, using a natural language program to increase spoken communication, and using matching-to-sample methods to teach categorization skills. We will record and review at least an hour of the ABA tutor's and parents' interactions with the child per week during unstructured and structured teaching situations. The purpose of these observations is to determine whether the parents are implementing the teaching strategies or behavior-management programs as designed (i.e., treatment integrity measures). If the ABA tutor or parent implements a program with less than 80% accuracy across two consecutive observations, an additional scripted role-play will be conducted as a booster session for the targeted skills.
  Arms: Technology-enhanced Early Intensive Behavioral Intervention
Behavioral: No-Intervention — The ABA tutors, parents/caregivers, and children will be randomly assigned to a wait-list control group.
  Arms: Wait-list No-intervention Control Group

SUMMARY:
The purpose of this study is to determine the extent to which technology may be used to provide (a) state-of-the-art assessment and intervention for children diagnosed with autism and (b) parent and tutor training for those who care for these children.

Children with autism often have problems with social interaction, language, and repetitive behavior (e.g., hand flapping and body rocking). Without early and intensive treatments, the long-term outcomes for children with autism are not very good; therefore, it is very important that effective treatments are started as soon as possible. Research has shown that Early Intensive Behavioral Interventions (EIBI) is an effective treatment for autism. Although EIBI is effective, most children with autism in military families do not receive EIBI because there are few professionals and paraprofessionals that are appropriately trained to do this, especially in the remote areas where military families tend to serve. The investigators want to show that web-based technologies (e.g., web-cams and internet-protocol cameras) can be used so that professionals in one place can treat children with autism anywhere in the world. The investigators also expect that providing these services will help children with autism improve their language, social, and academic skills. The investigators expect that the gains made by the children will help relieve many daily stressors and worries that families with children with autism have.

Children with autism who lack adaptive skills require constant help and supervision from parents. Thus, the improvements in the child's functioning will allow the child to become more independent and decrease parent stress associated with the need to constantly watch and help the child. Because EIBI services produce lasting improvements long after the intervention has ended, this project will provide both short-term and long-term benefits to the children who participate in the study, which will provide lasting relief to these dedicated military families.

In the long-term, this project may really change the way in which all (military and non-military) children and families get effective services that they cannot get now. Also, the results may help other professionals and researchers in psychology and medicine. That is, the results should be helpful to any kind of service that uses parent training and paraprofessionals. Most importantly, these services will improve the overall functioning of the children with autism and decrease the overall stress on these families as they continue to serve our country.

DETAILED DESCRIPTION:
1. Specific Aim: Technology-enhanced parent training. The investigators will assess whether E-Learning using the latest web-based instructional technologies provides an efficient and effective mechanism for training military parents of children with autism, regardless of their geographic location, to implement effective behavior management and teaching strategies with high procedural integrity (90% accuracy).

   - Hypothesis: Technology-enhanced parent training. Military parents who have a child with autism can be trained anywhere in the world to implement appropriate behavior management and teaching strategies based on the principles of applied behavior analysis (ABA) with 90% accuracy. Parents who receive this technology-enhanced training remotely will outperform those randomly assigned to a waitlist-control group on competency-based tests.
2. Specific Aim: Technology-enhanced ABA tutor training. The investigators will show that E-Learning using the latest web-based instructional technologies provides an efficient and effective mechanism for training adults to become ABA tutors who implement EIBI procedures with high procedural integrity (90% accuracy) in areas of the world where such services would otherwise be unavailable.

   - Hypothesis: Technology-enhanced ABA tutor training. Adults anywhere in the world with at least a high school diploma and no formal training in ABA can be trained in the basic principles of ABA and to implement EIBI therapy with 90% accuracy. Individuals who receive this technology-enhanced training remotely will outperform those randomly assigned to a waitlist-control group on both knowledge and competency-based tests.
3. Specific Aim: Technology-enhanced EIBI services. The investigators will demonstrate that technology-enhanced telehealth provides remote access to efficient and effective EIBI services to military families affected by autism.

   - Hypothesis: Technology-enhanced EIBI services. Young children with autism in military families who receive EIBI services that are supervised by University of Nebraska Medical Center (UNMC) experts remotely via technology-enhanced telehealth will show marked improvements in cognitive, language, social, play, and adaptive skills and decreases in problem behaviors relative to children randomly assigned to a wait-list control group.
4. Specific Aim: Reducing stress in military families affected by autism. The investigators will show that the provision of efficient and effective EIBI services using technology-enhanced telehealth will reduce family stress among military families affected by autism.

   * Hypothesis: Reducing stress in military families affected by autism. Military parents of children with autism who receive technology-enhanced EIBI services will show reductions in self-reported stress levels on both the Child Domain and Parent Domain subscales of the Parenting Stress Index relative to parents on the waitlist-control group.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion criteria for children with autism. a. Upon completion of the diagnostic assessment, children who meet the following inclusion criteria will be considered for participation. The inclusion criteria are:

   * (a) chronological age between 18 and 48 months of age,
   * (b) nonverbal mental age greater than 12 months (which is necessary to make an accurate diagnosis of autism in young children), and
   * (c) diagnosis of autism confirmed by meeting the cut-off scores on the autism diagnostic interview-revised (ADI-R) and the autism diagnostic observation schedule (ADOS)
2. Inclusion criteria for parents of children with autism. - All parents of children who are enrolled in this project will be invited to participate in Experiment 1 of this project if they are available for training during the course of the project.
3. Inclusion criteria for behavioral technicians.

   1. The participants for Experiment 2 will be young adults who are interested in being trained (at no cost) to provide ABA services to children with autism. Inclusion criteria for participation in this study are:

      * (a) age 19 or above;
      * (b) completion of, or enrollment in, an associate's or bachelor's degree program in psychology or a related field;
      * (c) completion of at least 12 semester credit hours at an accredited college or university;
      * (d) passage of criminal and abuse background checks; and (e) no prior training in ABA interventions.

Exclusion Criteria:

1. Exclusion criteria for children with autism

   a. Upon completion of the diagnostic assessment, children who meet the following exclusion criteria will be thanked for their participation, discharged from the project, and referred for services by other service providers. The exclusion criteria are:
   * (a) chronological age other than between 18 and 48 months of age,
   * (b) nonverbal mental age less than 12 months,
   * (c) no diagnosis of autism. In addition, children will be excluded if they have a serious medical condition that would interfere with treatment (e.g., blindness, deafness, cerebral palsy).
2. Exclusion criteria for parents of children with autism.

   a. Active duty military personnel who are unavailable due to deployment during this project will not participate, but will be offered parent training after their deployment is completed even if their data are not included in this project.
3. Exclusion criteria for behavioral technicians. a. Individuals who do not meet the inclusion criteria above and who cannot complete the physical requirements of the tasks involved in ABA therapy, which requires therapists to be able to speak, hear, see, sit, stand, walk, and lift 40 lbs. will be excluded from participation.

Ages: 18 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2012-05-30 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2018-07-01 (Estimated)

PRIMARY OUTCOMES:
Intelligent Quotient: Differential Abilities Scales, Second Edition | Time-to-Event Outcome Measure: Prior to and following intervention services (approximately 8 months)
  The investigators will use the Differential Abilities Scales, Second Edition (DAS-2; Elliott, 2007) as the primary dependent measure because it is particularly useful for measuring the cognitive abilities of young children; it covers a large age range (ages 2-6 to 17-11); it is well standardized; it has strong internal consistency and test-retest reliability (.90 to .95); and it correlates well with other measures of intelligence (M r = .76).

SECONDARY OUTCOMES:
Parent Training: Behavioral Implementation Skills for Play Activities | Time-to-Event Outcome Measure: Prior to and following parent-training curriculum (6 to 8 weeks)
  Almost all studies focusing on training parents and/or staff to implement behavior-analytic procedures include dependent measures that assess the extent to which parents display the following behaviors before and after training: (a) correct and incorrect instructions, (b) correct and incorrect prompts, (c) correct and incorrect consequences for appropriate behavior, and (d) correct and incorrect consequences for problem behavior. These basic measures can be adapted to measure procedural integrity.
Tutor Training: Behavioral Implementation of Work Activities | Time-to-Event Outcome Measure: Prior to and following tutor-training curriculum (9 to 12 weeks)
  Same dependent measure as described for the parent-training curriculum.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne W Fisher, Ph.D., Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States